CLINICAL TRIAL: NCT02461823
Title: The Influence of Porcelain Fused to Metal ( PFM) and Zirconia Crowns on Periodontal Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Ilan Hirsh MD, Senior staff Member Department of Periodontology, Rambam Health Care Campus, Haifa, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 078 -15-RMB CTIL
Record Dates: First submitted 2015-05-14; First posted 2015-06-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-05

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Z Crown (Experimental): A Zirconia crown will be provided to patients.
  Interventions: Device: Zirconia crown
- PFM Crown (Active Comparator): A Porcelain metal crown will provided to patients.
  Interventions: Device: Porcelain metal crown

INTERVENTIONS:
Device: Zirconia crown — patients will receive a Zirconia crown, the Zirconia crown will cover the natural crown.
  Arms: Z Crown
Device: Porcelain metal crown — patients will receive a porcelain fused to metal crown, the Porcelain metal crown will cover the natural crown.
  Arms: PFM Crown

SUMMARY:
Investigate the influence of the crown tye Porcelain fused to metal or Zirconia on periodontal health.

DETAILED DESCRIPTION:
Porcelain fused to metal (PFM) has been used in dentistry for the last five decades.

Zirconia (zirconium oxide, ZrO2) is the white crystalline powder oxide of the naturally occurring metal zirconium. Research of the medical utilization of zirconia dates back to the late 1960s. However, its utilization in dentistry did not start until the 1990s, when zirconia began to be used as a form of endodontic posts and implant abutments. The current literature contains studies that investigated the influence of zirconia implants and abutments on periodontal tissue, but to the investigators' knowledge, no work has been yet published which compares the influences of crown types on hard and soft tissues.

This prospective study will be conducted in the Department of Periodontology and in the Department of Maxillofacial Rehabilitation at Rambam Health Care Campus.

ELIGIBILITY:
inclusion criteria:

1. Patient age 18 - 85 years old
2. In need for one or more fixed partial prosthetic crown or bridge

exclusion criteria:

1. Smokers
2. Active periodontal disease
3. history of compromising systemic disease
4. Allergy to materials used in the study
5. current drug abuse
6. Pregnant or intend to become pregnant
7. severe salivary gland dysfunction
8. Severe medical complications ( organ transplants, cancer, immunocompromised, or undergoing long-term antibiotic or steroid therapy )

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
PgE2 ( Prostaglandin E2) | 4 months
  Gingival cervicular fluid samples will be attempt be planning Periotrom paper in the mesial and distal aspect of the experimental teeth.
  This samples will be assayed for PgE2 ( Prostaglandin E2) using Elyza kit. The concentration of PGE2 in gingival crevicular fluid will be examined around each tooth receiving a crown.

SECONDARY OUTCOMES:
PIaque index | 4 months
  The clinical examination will include measurement of PIaque index( soft tissue deposite around teeth)
GIingival index | 4 months
  The clinical examination will include measurement of the GIingival index (gingival inflamation around teeth)
Pocket depth | 4 months
  The clinical examination will include measurement of Pocket depth around teeth
Clinical attachment level | 4 months
  The clinical examination will include measurement of the Clinical attachment level around teeth
bone level | 4 months
  Periapical radiography will be obtain using customized film holding with Vinylpolysiloxan bite registration. Measurements of alveolar bone level will be performed on the digital images by a single examiner, using custom-made software.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ilan Hirsh, DMD, Principal Investigator — Rambam Health Care Campus , Department of Periodiontology, Haifa, Israel 31096